CLINICAL TRIAL: NCT03513952
Title: A Randomized Phase II Study of Atezolizumab (MPDL3280A) Plus Recombinant Human IL7 (CYT107) in Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: Atezolizumab and CYT107 in Treating Participants With Locally Advanced, Inoperable, or Metastatic Urothelial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-00684; NCI-2018-00684 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CITN-14 (Other: Cancer Immunotherapy Trials Network); CITN-14 (Other: CTEP); P30CA015704 (NIH); U01CA154967 (NIH)
Record Dates: First submitted 2018-05-01; First posted 2018-05-02 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-05

CONDITIONS: Advanced Bladder Urothelial Carcinoma; Advanced Ureter Urothelial Carcinoma; Metastatic Bladder Urothelial Carcinoma; Metastatic Renal Pelvis Urothelial Carcinoma; Metastatic Ureter Urothelial Carcinoma; Metastatic Urethral Urothelial Carcinoma; Metastatic Urothelial Carcinoma; Recurrent Bladder Urothelial Carcinoma; Recurrent Renal Pelvis Urothelial Carcinoma; Recurrent Ureter Urothelial Carcinoma; Recurrent Urethral Urothelial Carcinoma; Stage III Bladder Cancer AJCC v8; Stage III Renal Pelvis Cancer AJCC v8; Stage III Ureter Cancer AJCC v8; Stage III Urethral Cancer AJCC v8; Stage IV Bladder Cancer AJCC v8; Stage IV Renal Pelvis Cancer AJCC v8; Stage IV Ureter Cancer AJCC v8; Stage IV Urethral Cancer AJCC v8; Stage IVA Bladder Cancer AJCC v8; Stage IVB Bladder Cancer AJCC v8; Unresectable Bladder Urothelial Carcinoma; Unresectable Renal Pelvis Urothelial Carcinoma; Unresectable Ureter Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — atezolizumab; Biopsy; Specimen Handling; Interleukin-7; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (CYT107, atezolizumab) (Experimental): Patients receive CYT107 IM on days 1, 8, 15, and 22, and atezolizumab IV over 60 minutes on day 8 of cycle 1. Following cycle 1, patients receive atezolizumab IV over 30-60 minutes on day 1. Cycles with atezolizumab repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI scans, and collection of blood and stool samples on study. Patients may also undergo tumor biopsy at screening and on study.
  Interventions: Drug: Atezolizumab; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Glycosylated Recombinant Human Interleukin-7; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography and Computed Tomography Scan
- Group 2 (atezolizumab) (Active Comparator): Patients receive atezolizumab IV over 60 minutes on cycle 1. Following cycle 1, patients receive atezolizumab IV over 30-60 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI scans, and collection of blood and stool samples on study. Patients may also undergo tumor biopsy at screening and on study.
  Interventions: Drug: Atezolizumab; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography and Computed Tomography Scan
- Safety run in phase (Experimental): Patients assigned to the experimental arm (atezolizumab + CYT107). If the treatment combination of the experimental arm demonstrates an acceptable safety profile in the Safety Run-In (one or fewer patient experiences a protocol-defined Dose Limiting-Toxicity), randomized enrollment into the trial will begin. The Run-in phase patients will be analyzed and reported separately both for safety and for efficacy.
  Interventions: Drug: Atezolizumab; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Glycosylated Recombinant Human Interleukin-7; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography and Computed Tomography Scan

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Procedure: Biopsy — Undergo biopsy of tumor
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood and stool samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Glycosylated Recombinant Human Interleukin-7 — Given IM
  Other Names: CYT-107; CYT107; Glycosylated rhIL-7; INTERLEUKIN-7 HUMAN RECOMBINANT
  Arms: Group 1 (CYT107, atezolizumab); Safety run in phase
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography and Computed Tomography Scan — Undergo PET/CT
  Other Names: PET-CT Scan; PET/CT SCAN; Positron Emission Tomography/Computed Tomography

SUMMARY:
This phase II trial studies how well atezolizumab when given with glycosylated recombinant human interleukin-7 (CYT107) works in treating patients with urothelial carcinoma that has spread to nearby tissue or lymph nodes (locally advanced), cannot be removed by surgery (inoperable), or has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. CYT107 is a biological product naturally made by the body that may stimulate the immune system to destroy tumor cells. Giving atezolizumab and CYT107 may work better in treating patients with locally advanced, inoperable, or metastatic urothelial carcinoma compared to atezolizumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the clinical efficacy of the investigational treatment combination.

SECONDARY OBJECTIVES:

I. To determine the clinical activity and toxicity of the investigational treatment combination.

II. The clinical benefit rate (CBR), progression-free survival (PFS), duration of response (DOR), as measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune-related response criteria (irRC), and overall survival (OS).

III. The CBR, PFS, DOR, and OS in all patients and patients stratified by PD-L1 expression levels in the tumor microenvironment.

IV. The safety and toxicity of addition of CYT107 to atezolizumab.

EXPLORATORY OBJECTIVES:

I. To determine the immune correlates of the clinical activity of the investigational treatment combination.

II. Explore the effect of the investigational treatment combination on the number and phenotype of tumor-specific T cells in the peripheral blood.

III. Investigate for evidence that the investigational treatment combination increases the exposure of bladder cancer-specific antigens (e.g., cancer/testis antigens or neoantigens).

IV. Investigate changes in tumor microenvironment that correlate with response or provide information on potential actionable causes for lack of clinical benefit.

V. Investigate the potential that administration of atezolizumab with CYT107 may perturb the pharmacokinetics and immunogenicity of CYT107.

OUTLINE:

SAFETY RUN-IN PHASE: Patients assigned to the experimental arm (atezolizumab + CYT107). If the treatment combination of the experimental arm demonstrates an acceptable safety profile in the Safety Run-In (one or fewer patient experiences a protocol-defined Dose Limiting-Toxicity), randomized enrollment into the trial will begin. The Run-in phase patients will be analyzed and reported separately both for safety and for efficacy.

Patients are randomized to 1 of 2 groups.

GROUP 1 (experimental arm): Patients receive CYT107 intramuscularly (IM) on days 1, 8, 15, and 22, and atezolizumab intravenously (IV) over 60 minutes on day 8 of cycle 1. Following cycle 1, patients receive atezolizumab IV over 30-60 minutes on day 1. Cycles with atezolizumab repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) scans, and collection of blood and stool samples on study. Patients may also undergo tumor biopsy at screening and on study.

GROUP 2 (control arm): Patients receive atezolizumab IV over 60 minutes on cycle 1. Following cycle 1, patients receive atezolizumab IV over 30-60 minutes on day 1. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI scans, and collection of blood and stool samples on study. Patients may also undergo tumor biopsy at screening and on study.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented locally advanced/inoperable or metastatic urothelial bladder carcinoma (UBC), including renal pelvis, ureters, urinary bladder, and urethra

  * Note: Mixed histology tumors allowed if predominant histology is urothelial carcinoma
  * Note: Small cell or neuroendocrine carcinoma is not allowed if predominant
* Patients must have recurrent disease after any prior platinum-based chemotherapy regimen
* Patients must have measurable disease per RECIST 1.1 assessed by computed tomography (CT) scan or magnetic resonance imaging (MRI)
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Patients must have a life expectancy of greater or equal to 12 weeks
* Leukocytes >= 2,500/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert's disease who have serum bilirubin level =< 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN (AST and/or ALT=< 5 x ULN for patients with liver involvement)
* Alkaline phosphatase =< 2.5 x ULN (=< 5 x ULN for patients with documented liver involvement or bone metastases)
* Creatinine clearance >= 30 mL/min/1.73 m^2 by Cockcroft-Gault

  * At the discretion of the treating physician, a 24-hour urine creatinine clearance could be obtained and utilized as the gold standard if creatinine clearance by Cockcroft-Gault is < 30, and prevents patient enrollment on the trial
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose)
* Patients must provide tissue from an archival tumor sample (obtained within 2 years from screening visit) or newly obtained core, punch, or excisional biopsy of a tumor lesion if deemed relatively safe and technically feasible
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours before receiving the first dose of study agent(s); if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;

  * Administration of atezolizumab may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality; CYT107 has not been tested for reproductive toxicity yet and may expose to the same risk; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) before study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of study agent; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* Patients positive for human immunodeficiency virus (HIV) are allowed on study, but HIV-positive patients must have:

  * A stable regimen of highly active antiretroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard polymerase chain reaction (PCR)-based tests

Exclusion Criteria:

* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Patients who have had chemotherapy or radiotherapy within 2 weeks (4 weeks for nitrosoureas or systemic mitomycin C) before the initiation of study treatment
* Patients who have received more than 2 systemic cytotoxic chemotherapy regimens for metastatic urothelial carcinoma

  * Note: Prior perioperative chemotherapy is allowed and is not counted as a line of therapy if patient relapsed >= 12 months later and received additional platinum-based chemotherapy for metastatic disease
* Patients who have not recovered from adverse events (other than alopecia) due to agents administered more than 4 weeks earlier (i.e., have residual toxicities > grade 1); however, the following therapies are allowed:

  * Hormone-replacement therapy or oral contraceptives
  * Herbal therapy >= 1 week before initiation of study treatment (herbal therapy intended as anticancer therapy must be discontinued at least 1 week before initiation of study treatment)
  * Palliative radiotherapy for bone metastases > 2 weeks before initiation of study treatment
* Patients who have received prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody, or pathway -targeting agents

  * Patients who have received prior treatment with anti-CTLA-4 may be enrolled, provided the following requirements are met:

    * Minimum of 12 weeks from the first dose of anti-CTLA-4 and > 6 weeks from the last dose
    * No history of severe immune-related adverse effects from anti-CTLA-4 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] grade 3 and 4)
* Patients who have received treatment with any other investigational agent within 4 weeks before initiation of study treatment
* Patients who have received treatment with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2) within 6 weeks before initiation of study treatment
* Patients who have received treatment with systemic immunosuppressive medications (including, but not limited to, oral prednisone ( > 10 mg/day or equivalent), cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti TNF] agents) within 2 weeks before initiation of study treatment

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
  * The use of inhaled corticosteroids, and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Patients taking bisphosphonate therapy for symptomatic hypercalcemia

  * Note: Use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed
* Patients with known primary central nervous system (CNS) malignancy or symptomatic CNS metastases are excluded, with the following exceptions:

  * Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

    * Evaluable or measurable disease outside the CNS
    * No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
    * No history of intracranial hemorrhage or spinal cord hemorrhage
    * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted
    * No neurosurgical resection or brain biopsy within 28 days before initiation of study treatment
  * Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

    * Radiographic demonstration of improvement upon the completion of CNS directed therapy and no evidence of interim progression between the completion of CNS directed therapy and the screening radiographic study
    * No stereotactic radiation or whole-brain radiation within 28 days before initiation of study treatment
    * Screening CNS radiographic study >= 4 weeks from completion of radiotherapy and >= 2 weeks from discontinuation of corticosteroids
  * Note: Patients with CNS metastases enrolled on trial must also have a brain MRI imaging at all standard radiologic evaluation timepoints
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Patients who have a history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients with known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver/nonalcoholic fatty liver disease (NAFLD)/nonalcoholic steatohepatitis (NASH); and inherited liver disease

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Patients with active underlying autoimmune disease requiring systemic immunosuppressive medication (oral prednisone > 10 mg/day or equivalent). Topical, inhaled, or intra-articular steroids or physiologic endocrine replacement (insulin, levothyroxine, etc.) are permitted. Patients with a history of autoimmune disease that is not currently active require consultation with the protocol principal investigator (PI) and/or Cancer Immunotherapy Trials Network (CITN) Coordinating Center
* Patients who have a history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Patients who have known additional malignancies other than UBC within 2 years before initiation of study treatment; exceptions include malignancies with a negligible risk of metastasis or death and treated with expected curative outcome (e.g., non-melanomatous skin cancers), or localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer
* Patients with active tuberculosis (TB)
* Patients who have leptomeningeal disease
* Patients who have severe infections within 4 weeks before initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia;

  * Exception: Uncomplicated urinary tract infection will not be considered as a severe infection in these patients
* Patients who have signs or symptoms of infection within 2 weeks before initiation of study treatment
* Patients who have received oral or IV antibiotics within 2 weeks before initiation of study treatment; patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Patients who have major surgical procedure, other than for diagnosis, within 28 days before initiation of study treatment or anticipation of need for a major surgical procedure during the course of the study
* Patients who have had a live, attenuated vaccine within 4 weeks before initiation of study treatment or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab.

  * Influenza vaccination should be given during influenza season only (approximately October to March); patients must not receive live, attenuated influenza vaccine within 4 weeks before initiation of study treatment or at any time during the study
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure (New York Heart Association class III or IV), unstable angina pectoris, cardiac arrhythmia, recent myocardial infarction (within the last 6 months), or psychiatric illness/social situations that would limit compliance with study requirements
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or medical (e.g., infectious) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Y Yu, Principal Investigator — Cancer Immunotherapy Trials Network
Locations (9):
- United States (9):
  - Kaiser Permanente-Riverside, Riverside, California
  - Moffitt Cancer Center, Tampa, Florida
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - East Jefferson General Hospital, Metairie, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - FHCC South Lake Union, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety Run-In Phase: If the treatment combination demonstrates an acceptable safety profile (one or fewer patient experiences a protocol-defined Dose Limiting-Toxicity), randomized enrollment will begin.
Groups:
- Group 1 (CYT107, Atezolizumab): Patients receive CYT107 on days 1, 8, 15, and 22, and atezolizumab on day 8 of cycle 1. Following cycle 1, patients receive atezolizumab on day 1. Cycles with atezolizumab repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Atezolizumab: Given IV
  Glycosylated Recombinant Human Interleukin-7: Given IM
- Group 2 (Atezolizumab): Patients receive atezolizumab on Day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Atezolizumab: Given IV
- Safety Run in Phase: Patients were not randomized; they were assigned to the experimental arm treatment (atezolizumab + CYT107). Patients receive CYT107 on days 1, 8, 15, and 22, and atezolizumab on day 8 of cycle 1. Following cycle 1, patients receive atezolizumab on day 1. Cycles with atezolizumab repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Atezolizumab: Given IV
  Glycosylated Recombinant Human Interleukin-7: Given IM
Period: Overall Study
Arm/Group | Group 1 (CYT107, Atezolizumab) | Group 2 (Atezolizumab) | Safety Run in Phase
Started | 19 | 21 | 7
Completed (Completed Study Treatment (up to 2 years)) | 3 | 2 | 0
Not Completed | 16 | 19 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (CYT107, Atezolizumab) | Group 2 (Atezolizumab) | Safety Run in Phase | Total
Number analyzed (Participants) | 19 | 21 | 7 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (9.2) | 66.3 (8.5) | 59.7 (11) | 65.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 1 | 9
  Male | 16 | 16 | 6 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 19 | 19 | 6 | 44
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 3
  White | 19 | 18 | 7 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 21 | 7 | 47

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the proportion of patients who have achieved Complete Response (CR) - disappearance of all target lesions or Partial Response (PR) - >=30% decrease in the sum of the longest diameter of target lesions according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (CYT107, Atezolizumab) | Group 2 (Atezolizumab) | Safety Run in Phase
Number analyzed (Participants) | 19 | 21 | 7
Participants
  Partial Response (PR) | 3 | 4 | 0
  Complete Response (CR) | 2 | 1 | 0
  Combined total PR + CR | 5 | 5 | 0
Statistical Analysis 1: Comparison: Group 1 (CYT107, Atezolizumab) vs Group 2 (Atezolizumab); Test type: Superiority; p = 0.428, Cochran-Mantel-Haenszel — A one-sided significance level of 0.10 will be considered for the test; Estimations were done separately in each treatment arm; the difference between treatments was not calculated

2. Secondary Outcome: Clinical Benefit Rate (CBR) Measured by RECIST v1.1
Description: CBR is defined as the percentage of patients with advanced or metastatic cancer who have achieved CR (disappearance of all target lesions), PR (>=30% decrease in the sum of the longest diameter of target lesions), and stable disease (SD) (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum diameters of target lesions) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1; CBR = CR + PR + SD.
  Will also assess CBR in patients stratified by PD-L1 expression levels in the tumor microenvironment.
Time Frame: Up to 2 years
Population: The PD-L1 assay produced no data due to expired antibody. Stratification by PD-L1 expression levels in the tumor microenvironment cannot be reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (CYT107, Atezolizumab) | Group 2 (Atezolizumab) | Safety Run in Phase
Number analyzed (Participants) | 19 | 21 | 7
Participants
  Stable Disease (SD) | 2 | 4 | 2
  Partial Response (PR) | 3 | 4 | 0
  Complete Response (CR) | 2 | 1 | 0
  Combined total CR + PR + SD | 7 | 9 | 2
Statistical Analysis 1: Comparison: Group 1 (CYT107, Atezolizumab) vs Group 2 (Atezolizumab); Test type: Equivalence — Two-sided Cochran-Mantel-Haenszel test for the CBR was performed, which is used for testing zero effect or "equivalence" between treatments. A two-sided significance level of 0.05 will be considered for the test; p = 0.702, Cochran-Mantel-Haenszel; Risk Difference (RD) = -6.0, 95% CI 2-sided [-36.3 to 24.3]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression is defined, per RECIST v1.1, as a 20% increase in the sum of the longest diameter of target lesions (the sum must demonstrate an absolute increase of at least 5 mm), or the appearance of new lesions and/or unequivocal progression of non-target lesions.
  PFS will be summarized using Kaplan-Meier estimates. Will also assess PFS in patients stratified by PD-L1 expression levels in the tumor microenvironment.
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 2 years.
Population: Patients without documented PD or death are censored at the last disease assessment date.
  The PD-L1 assay produced no data due to expired antibody. Stratification by PD-L1 expression levels in the tumor microenvironment cannot be reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 (CYT107, Atezolizumab) | Group 2 (Atezolizumab) | Safety Run in Phase
Number analyzed (Participants) | 19 | 21 | 7
months | 2.1 [1.2 to 6.1] | 2.2 [1.8 to 4.6] | 2.1 [1.1 to 4.0]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is measured by RECIST v1.1. DOR will be summarized using Kaplan-Meier estimates. Will also assess DOR in patients stratified by PD-L1 expression levels in the tumor microenvironment.
Time Frame: Time interval between the date of first response (CR/PR) and the date of progression, assessed up to 2 years.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 (CYT107, Atezolizumab) | Group 2 (Atezolizumab) | Safety Run in Phase
Number analyzed (Participants) | 19 | 21 | 0
months | NA [2.3 to NA] — The medians and 95% CIs for DOR were calculated based on Kaplan-Meier estimates. The Kaplan-Meier curve does not cross the 50% probability; therefore, the median survival time could not be calculated. Insufficient events to calculate a reliable upper 95% CI. | NA [4.0 to NA] — The medians and 95% CIs for DOR were calculated based on Kaplan-Meier estimates. The Kaplan-Meier curve does not cross the 50% probability; therefore, the median survival time could not be calculated. Insufficient events to calculate a reliable upper 95% CI. |

5. Secondary Outcome: Overall Survival (OS)
Description: OS will be summarized using Kaplan-Meier estimates. Will also assess OS in patients stratified by PD-L1 expression levels in the tumor microenvironment.
Time Frame: Time interval between start of treatment to death due to any cause, assessed up to 48 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 (CYT107, Atezolizumab) | Group 2 (Atezolizumab) | Safety Run in Phase
Number analyzed (Participants) | 19 | 19 | 7
months | 9.1 [2.6 to NA] — The medians and 95% CIs for OS were calculated based on Kaplan-Meier estimates. Insufficient events to calculate a reliable upper 95% CI. | 10.4 [4.7 to 20.7] | 4.5 [1.1 to 9.8]

6. Other Pre Specified Outcome: Assessment of Investigation Treatment Combination on the Immune-bias of the Tumor Microenvironment
Description: The evaluation of the effect of the investigation treatment combination on the immune-bias of the tumor microenvironment, based upon baseline and post-baseline tumor biopsy comparisons of number, distribution, and phenotype of tumor-infiltrating cells; PD-L1 expression, and expression of Interferon gamma (IFN-gamma) and associated proinflammatory gene expression in the tumor microenvironment.
Time Frame: Up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and other (not including serious) adverse events were assessed for up to 30 days post-treatment. All-cause mortality was assessed for up to 48 months.
Description: Two patients randomized in Group 2 (Atezolizumab) did not receive any study treatment, therefore the total number of participants at risk in the Serious Adverse Events and other (not including serious) adverse events tables were adjusted accordingly.
Arm/Group | Group 1 (CYT107, Atezolizumab) | Group 2 (Atezolizumab) | Safety Run in Phase
All-Cause Mortality (participants affected / at risk) | 11/19 | 14/21 | 6/7
Serious Adverse Events (participants affected / at risk) | 13/19 | 11/19 | 5/7
Other Adverse Events (participants affected / at risk) | 18/19 | 19/19 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (CYT107, Atezolizumab) (N=19) | Group 2 (Atezolizumab) (N=19) | Safety Run in Phase (N=7)
Anemia (Blood and lymphatic system disorders) | 1 | 3 | 1
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Esophageal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Death NOS (General disorders) | 1 | 0 | 0
Disease Progression (General disorders) | 1 | 0 | 1
Edema Limbs (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Fever (General disorders) | 0 | 1 | 1
Generalized Edema (General disorders) | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 1 | 0
Lung Infection (Infections and infestations) | 1 | 1 | 1
Sepsis (Infections and infestations) | 2 | 1 | 1
Upper Respiratory Infection (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 1
Creatinine Increased (Investigations) | 2 | 0 | 0
Lipase Increased (Investigations) | 0 | 1 | 0
Serum Amylase Increased (Investigations) | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Concentration Impairment (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1 | 0
Stroke (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 3 | 0
Acute Tubular Necrosis (Renal and urinary disorders) | 0 | 1 | 0
Cystitis Noninfective (Renal and urinary disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 2 | 2 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urosepsis (Renal and urinary disorders) | 1 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0
Thromboembolic Event (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (CYT107, Atezolizumab) (N=19) | Group 2 (Atezolizumab) (N=19) | Safety Run in Phase (N=7)
Anemia (Blood and lymphatic system disorders) | 7 | 8 | 3
DVT (Blood and lymphatic system disorders) | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 2 | 0
Hypervolemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Chest Pain - Cardiac (Cardiac disorders) | 0 | 1 | 0
Diastolic Dysfunction (Cardiac disorders) | 0 | 1 | 0
Heart Failure (Cardiac disorders) | 0 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 2 | 0
Sinus Tachycardia (Cardiac disorders) | 3 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1
Right Ear Impaction (Ear and labyrinth disorders) | 0 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Blurred Vision (Eye disorders) | 1 | 0 | 0
Floaters (Eye disorders) | 0 | 1 | 0
Itchy Eyes (Eye disorders) | 1 | 0 | 0
Tunnel Vision (Eye disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 7 | 0
Anal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 0
Colonic Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 8 | 6 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 8 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Esophageal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Fecal Incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 3 | 4
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 4
Bilateral Pulmonary Emboli (General disorders) | 0 | 1 | 0
Chills (General disorders) | 4 | 0 | 2
DVT (General disorders) | 1 | 0 | 0
Edema Limbs (General disorders) | 2 | 1 | 1
Fatigue (General disorders) | 11 | 8 | 3
Fever (General disorders) | 4 | 2 | 3
Generalized Edema (General disorders) | 1 | 0 | 0
Hydronephrosis (General disorders) | 0 | 1 | 0
Hypochloremia (General disorders) | 1 | 0 | 0
Increased Prothrombin (General disorders) | 1 | 0 | 0
Injection Site Reaction (General disorders) | 1 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 1 | 1
Pain (General disorders) | 3 | 2 | 1
Physical Deconditioning (General disorders) | 0 | 1 | 0
Redness at Injection Site (General disorders) | 0 | 1 | 0
Shaking/Shivering (General disorders) | 0 | 0 | 1
Swelling at Injection Site (General disorders) | 1 | 0 | 0
Abdominal Infection (Infections and infestations) | 1 | 0 | 0
Autoimmune Hepatitis (Infections and infestations) | 1 | 0 | 0
Covid (Infections and infestations) | 0 | 1 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 0
Tooth Infection (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 3 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 4 | 1 | 1
Alkaline Phosphatase Increased (Investigations) | 6 | 3 | 3
aPTT Decreased (Investigations) | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 4 | 2 | 2
Blood Bilirubin Increased (Investigations) | 1 | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 2 | 2 | 0
BUN Increased (Investigations) | 0 | 1 | 0
CD4 Lymphocytes Decreased (Investigations) | 0 | 1 | 0
CD8 Lymphocytes Decreased (Investigations) | 0 | 1 | 0
Creatinine Increased (Investigations) | 9 | 6 | 3
Elevated BUN (Investigations) | 0 | 2 | 0
Hemoglobin Increased (Investigations) | 0 | 1 | 0
Hypochloremia (Investigations) | 0 | 1 | 0
Increased BUN (Investigations) | 1 | 0 | 0
INR Increased (Investigations) | 1 | 4 | 0
Lactic Acid Increased (Investigations) | 0 | 1 | 0
LDH Increased (Investigations) | 1 | 1 | 0
Lipase Increased (Investigations) | 0 | 1 | 0
Lymphocyte Count Decreased (Investigations) | 3 | 4 | 0
Lymphocyte Count Increased (Investigations) | 1 | 0 | 0
Monocytosis (Investigations) | 0 | 1 | 0
Neutrophil Count Decreased (Investigations) | 2 | 2 | 0
Neutrophilia (Investigations) | 1 | 1 | 0
Platelet Count Decreased (Investigations) | 2 | 5 | 0
Prolonged Prothrombin Time (Investigations) | 0 | 1 | 0
Shoulder Pain (Investigations) | 0 | 1 | 0
Thrombocytosis (Investigations) | 1 | 0 | 0
Thyroid Stimulating Hormone Increased (Investigations) | 1 | 0 | 0
Total Protein Elevated (Investigations) | 0 | 1 | 0
WBC Increased (Investigations) | 1 | 0 | 0
Weight Loss (Investigations) | 2 | 0 | 0
White Blood Cell Decreased (Investigations) | 1 | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 5 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 5 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 4 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 7 | 7 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Rotator Cuff Injury (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Trigger Finger, Left Hand (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Brain Mets (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 1
Dysgeusia (Nervous system disorders) | 2 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 6 | 1 | 0
Memory Impairment (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1 | 1
Spasticity (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1
Confusion (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Distracted and Forgetful (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1 | 0
Bladder Spasm (Renal and urinary disorders) | 1 | 0 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 3 | 1 | 0
Hydroneprosis (Renal and urinary disorders) | 1 | 0 | 0
Nephrostomy Dislodgment (Renal and urinary disorders) | 1 | 0 | 0
Nocturia - Intermittent (Renal and urinary disorders) | 1 | 0 | 0
Renal Injury (Renal and urinary disorders) | 1 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 2 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 2 | 0 | 1
Urinary Urgency (Renal and urinary disorders) | 0 | 1 | 0
Urine Discoloration (Renal and urinary disorders) | 1 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 2 | 0 | 0
Perineal Pain (Reproductive system and breast disorders) | 1 | 0 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Itching and Discomfort Around Ostomy/Stoma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ostomy/Stome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Possible Folliculitis/Rash Around Stoma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2 | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4 | 3 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Slight Itch All Over Body (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Stoma/Ostomy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Sun Burn Blisters (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Suspicious for SCC (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Tissue Sloughing (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 4 | 2
Hypotension (Vascular disorders) | 4 | 2 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 0
Thromboembolic Event (Vascular disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT03513952/Prot_SAP_000.pdf